CLINICAL TRIAL: NCT01485237
Title: Severe Pandemic H1N1 Infection in ICU: Comparative Resource Utilization
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Dr. Anand Kumar, Intensivist, University of Manitoba
Other Study IDs: pandemic001; H2009:175 (Other: University of Manitoba Research Ethics Board Identifier:)
Record Dates: First submitted 2011-12-01; First posted 2011-12-05 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Novel H1N1 Influenzal Acute Respiratory Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Severe H1N1 pneumonia in adult patients: Severe adult H1N1 pneumonia patients undergoing antiviral and oxygen therapy, mechanical ventilation and support with pulmonary rescue therapies ( nitric oxide, ECMO, HFO)in Winnipeg
  Interventions: Other: We will compare the resources used by both groups
- Severe pneumonia in adults not H1N1: Patients admitted to the hospital and/or ICU with viral pneumonia, bacterial pneumonia, septic shock, ARDS in Winnipeg
  Interventions: Other: We will compare the resources used by both groups

INTERVENTIONS:
Other: We will compare the resources used by both groups — The main purpose of this study is to review the resource utilization. Secondary objectives include, comparison of resource utilization to other similar disorders (viral pneumonia, bacterial pneumonia, septic shock, ARDS). We will also look at the percentage of patients that required ICU care as compared to those who could be cared for on medical wards. We will determine the resources used by both groups and compare. Finally we will record the frequency of chronic comorbidities in hospitalized adult H1N1 patients.

SUMMARY:
The main purpose of this study is to review the resource utilization of severe adult H1N1 pneumonia undergoing antiviral and oxygen therapy, mechanical ventilation and support with pulmonary rescue therapies ( nitric oxide, ECMO, HFO) in critically ill patients in Winnipeg. Secondary objectives include, comparison of resource utilization to other similar disorders (viral pneumonia, bacterial pneumonia, septic shock, ARDS). The investigators will also look at the percentage of patients that required ICU care as compared to those who could be cared for on medical wards. The investigators will determine the resources used by both groups and compare. Finally the investigators will record the frequency of chronic comorbidities in hospitalized adult H1N1 patients.

ELIGIBILITY:
Inclusion Criteria:

1. > 18years,
2. Suspected or confirmed influenza (Appendix A)
3. Requirement for ICU admission due to respiratory distress or critical illness defined as one of:a) Inspired oxygen need of >50% for at least 4 hours (For FiO2 for non-intubated patients see Appendix B) b) mechanical ventilation c) Patient is receiving inotrope or vasopressor

Exclusion Criteria:

1. Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe adult H1N1 pneumonia undergoing antiviral and oxygen therapy, mechanical ventilation and support with pulmonary rescue therapies ( nitric oxide, ECMO, HFO) in critically ill patients in Winnipeg. Patients with other similar disorders (viral pneumonia, bacterial pneumonia, septic shock, ARDS)that may require some of the same treatments.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anand Kumar, MD, Principal Investigator — Health Sciences Centre, Winnipeg
Locations (1):
- Health Sciences Centre, Winnipeg, Winnipeg, Manitoba, Canada